CLINICAL TRIAL: NCT04217252
Title: Clinical Application of High-throughput Sequencing Technology for the Diagnosis of Patients With Severe Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the impact of the COVID-19, the project has been suspended for a long time and cannot continue to complete.
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Lingxiao Jiang, Senior Technologist, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20191230
Record Dates: First submitted 2019-12-30; First posted 2020-01-03 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Infection
Keywords: severe infection; high throughput sequencing; infectious pathogen
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: The participants from the department of hematology and intensive care unit who meet the inclusion criteria are randomly divided into the control group and the experimental group. Both the participants of the control group and the experimental group undergo routine clinical diagnosis methods and treatment. In addition, the participants of the experimental group are collected the samples including whole blood, cerebrospinal fluid or alveolar lavage fluid required for high throughput sequencing of infectious pathogens during sample collection for routine pathogenic examination of infection.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental): high throughput sequencing of infectious pathogens
  Interventions: Diagnostic Test: PMseqTM high-throughput sequencing technology
- the control group (No Intervention): no intervention

INTERVENTIONS:
Diagnostic Test: PMseqTM high-throughput sequencing technology — high throughput sequencing of infectious pathogens
  Arms: the experimental group

SUMMARY:
The purpose of this study is to evaluate the clinical value of high throughput sequencing of infectious pathogens for patients with severe infection, and to establish foundation for high throughput sequencing to be the clinical routine infection pathogen examination. This study is a diagnostic study, and the sample size is 320 cases. 320 participants from the department of hematology and intensive care unit who meet the inclusion criteria are randomly divided into the control group and the experimental group with 160 cases in each group. Both the participants of the control group and the experimental group undergo routine clinical diagnosis methods and treatment. In addition, the participants of the experimental group are collected the samples including whole blood, cerebrospinal fluid or alveolar lavage fluid required for high throughput sequencing of infectious pathogens during sample collection for routine pathogenic examination of infection. The pathogen diagnosis rate and the diagnostic accuracy rate between the conventional infectious pathogen tests and the high throughput sequencing of infectious pathogens will be compared in the experimental group. By gathering statistics of consultation hours and cost efficiency, the effect of high throughput sequencing of infectious pathogens on the diagnosis and treatment efficiency of the experimental group and the control group will be compared, and through these indicators, clinical application value for the diagnosis of severe infection patients by high throughput sequencing of infectious pathogens can be evaluated.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical value of high throughput sequencing of infectious pathogens for patients with severe infection, and to establish foundation for high throughput sequencing to be the clinical routine infection pathogen examination.

This study is a diagnostic study, and the sample size is 320 cases. 320 participants from the department of hematology and intensive care unit who meet the inclusion criteria are randomly divided into the control group and the experimental group with 160 cases in each group. Both the participants of the control group and the experimental group undergo routine clinical diagnosis methods and treatment. In addition, the participants of the experimental group are collected the samples including whole blood, cerebrospinal fluid or alveolar lavage fluid required for high throughput sequencing of infectious pathogens during sample collection for routine pathogenic examination of infection. For the experimental group participants, the clinicians will comprehensively determine the follow-up diagnosis methods and treatment according to the clinical routine infection pathogen tests results combining with the results of high throughput sequencing of infectious pathogen, while the control group participants proceed to undergo follow-up diagnosis methods and treatment according to the results of the clinical routine infection pathogen examination. If the results of high throughput sequencing of infectious pathogens of the test group are inconsistent with the results of clinical routine infection pathogen examination, the follow-up diagnosis and treatment of the participants will be based on the results of clinical routine infection pathogen examination with priority.

For sample size assessment, we have predicted the pathogen diagnosis rate of routine clinical pathogen detection methods and high-throughput sequencing of infectious pathogens (α=0.05, β=0.10 (power=0.9)), considering that the maximum rate of missing cases was 20%, and finally got the sample content. And this study will include all subjects selected and randomized into a full analysis set under the intent-to-treat principle. After excluding participants with insufficient sample, withdrawing from the trial midway, giving up treatment and leaving the hospital, or lost to follow-up, the remaining participants will be included in the protocol set under the per-protocol principle.

As for statistical analysis, the pathogen diagnosis rate and the diagnostic accuracy rate between the conventional infectious pathogen tests and the high throughput sequencing of infectious pathogens will be compared in the experimental group. By gathering statistics of consultation hours and cost efficiency, the effect of high throughput sequencing of infectious pathogens on the diagnosis and treatment efficiency of the experimental group and the control group will be compared, and through these indicators, clinical application value for the diagnosis of severe infection patients by high throughput sequencing of infectious pathogens can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 years old, male or female
* Body temperature > 38 ℃
* Newly admitted patients
* The clinician judges that the patient may be infected, and need to undergo the infection pathogen tests
* The patients volunteer to participate in this study and sign informed consent form

Exclusion Criteria:

* Those who do not meet the inclusion criteria
* The patients who can't cooperate

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
pathogen diagnosis rate | through study completion, an average of half a year
  probability of pathogens detected
the diagnostic accuracy rate | through study completion, an average of half a year
  probability of diagnosing correctly for high throughput sequencing of infectious pathogen

SECONDARY OUTCOMES:
money spent by participant | through study completion, an average of half a year
  the money the participant spent during hospitalization
consultation hours | through study completion, an average of half a year
  time of diagnosis and treatment for the participant

OTHER OUTCOMES:
the amount and type of antibiotics used | through study completion, an average of half a year
  the amount and type of antibiotics used by participants in the hospital for diagnosis and treatment
28-day mortality | through study completion, an average of half a year
  participants mortality within 28 days
in-hospital mortality | through study completion, an average of half a year
  participants mortality during hospitalization
anti-infective treatment time | through study completion, an average of half a year
  the time using for treating infection
the time with effective body temperature control | through study completion, an average of half a year
  the time that body temperature of a participant is effectively and continuously controlled

CONTACTS AND LOCATIONS:
Overall Officials: Lingxiao Jiang, Principal Investigator — Division of Laboratory Medicine, Zhujiang Hospital

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP
Time Frame: starting 1 year after publication
Access Criteria: Related researchers